CLINICAL TRIAL: NCT07176559
Title: Pilot Randomized Clinical Trial of Informational Support Versus Spiritual Care
Acronym: PRaCTIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: The Walther Cancer Foundation (Unknown)
Responsible Party: Principal Investigator, Alexia M. Torke, Professor of Medicine and Section Chief, Palliative Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IUSCCC-0936
Record Dates: First submitted 2025-08-29; First posted 2025-09-16 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Stage IV Lung Cancer; Lung Cancer; Gastrointestinal Malignancy
Keywords: lung cancer; gastrointestinal cancer; spiritual care; spiritual wellbeing; spirituality
MeSH Terms: conditions — Lung Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chaplain Intervention Group (Experimental): Eligible and consented participants that are randomized to the Chaplain Intervention Group will receive a total of 4 visits with a board-certified or board-eligible chaplain. These visits will occur weekly for approximately 4 weeks either in person, by telephone, or through a HIPAA compliant video platform. The visits will last an average of 30 minutes each.
  Interventions: Behavioral: Chaplain Intervention Group
- Attention Control Group (No Intervention): Eligible and consented patients randomized to the Attention Control group will receive 4 visits with a trained social worker. The visits will be conducted weekly for approximately 4 weeks. Each visit will take place for approximately 30 minutes.

INTERVENTIONS:
Behavioral: Chaplain Intervention Group — Eligible and consented participants that are randomized to the Chaplain Intervention Group will receive a total of 4 visits with a board-certified or board-eligible chaplain. These visits will occur weekly for approximately 4 weeks either in person, by telephone, or through a HIPAA compliant video platform. The visits will last an average of 30 minutes each.
  Arms: Chaplain Intervention Group

SUMMARY:
The purpose of this study is to address the need for effective spiritual care support for patients with lung and gastrointestinal cancer. This study will examine how spiritual care affects spiritual wellbeing, anxiety, depression, satisfaction with spiritual care, and quality of communication.

DETAILED DESCRIPTION:
This study is an individually randomized trial of chaplain-led intervention utilizing the Spiritual Care Assessment and Intervention (SCAI) framework compared to attention control. The chaplain intervention will consist of 4 spiritual care visits with a board-certified or board-eligible chaplain once a week for approximately 4 weeks. The attention control group will consist of 4 study visits with a trained social worker once a week for approximately 4 weeks.

Participants will be randomized 1:1 to the chaplain or attention control group.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Ability to provide informed consent and HIPAA authorization
3. Subject is at least 2 weeks post-diagnosis of an incurable and advanced stage (IV) lung or gastrointestinal (GI) malignancy and receiving cancer care at IU Simon Cancer Center, other IU Health Oncology Clinics, or Eskenazi Health Oncology Clinics
4. Subject has a reliable phone and is willing to participate in 4 sessions with the chaplain
5. ECOG score ranging from 0 (fully active) to 3 (able to conduct limited self-care in bed or chair more than 50% of waking hours)
6. Has low Spiritual Well-Being score of 35 or less on the FACIT-Sp
7. Subject makes 2 or fewer errors on the Callahan 6-item cognitive screener administered during screening

Exclusion Criteria:

1. Subject makes 3 or more errors on the Callahan 6-item cognitive screener administered during screening, or exhibits significant psychiatric or cognitive impairment (e.g., dementia/delirium, intellectual disability, active psychosis) that in the judgment of the research team would preclude providing informed consent and study participation
2. Currently receiving hospice care Note: subjects who enroll in hospice during the trial will have the option of continuing trial participation
3. Have had a visit with a healthcare chaplain within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of feasibility of the Spiritual Care Assessment and Intervention (SCAI) framework vs the attention control group | Weekly visits 1-4, within 3 months of enrollment
  Percentage of participants completing interviews
Evaluation of acceptability of the Spiritual Care Assessment and Intervention (SCAI) framework vs the attention control group | Weekly visits 1-4, within 3 months of enrollment
  Acceptability Intervention Measure and Treatment Acceptability and Adherence Scales
Test the effects of spiritual care on the outcome of spiritual wellbeing | Baseline, 1, 6, and 12 weeks post intervention
  Measured by the Functional Assessment of Chronic Illness Therapy - Spirituality

SECONDARY OUTCOMES:
Effects of Spiritual Care Assessment and Intervention (SCAI) framework on anxiety with spiritual care | 1, 6, and 12 weeks post intervention
  Generalize Anxiety Disorder - 7
Effects of Spiritual Care Assessment and Intervention (SCAI) framework on depression with spiritual care | 1, 6, and 12 weeks post intervention
  Patient Health Questionnaire-8
Effects of Spiritual Care Assessment and Intervention (SCAI) framework on satisfaction with spiritual care | 1, 6, and 12 weeks post intervention
  Patient Satisfaction Instrument-Chaplaincy and Client Satisfaction Questionnaire
Effects of Spiritual Care Assessment and Intervention (SCAI) framework on spirituality | 1, 6, and 12 weeks post intervention
  Patient-Reported Outcomes Measurement Information System 7
Effects of Spiritual Care Assessment and Intervention (SCAI) framework on religious coping | 1, 6, and 12 weeks post intervention
  Brief Religious Coping Scale (RCOPE)
Effects of Spiritual Care Assessment and Intervention (SCAI) framework on positive affect | 1, 6, and 12 weeks post intervention
  Patient-Reported Outcomes Measurement Information System (PROMIS) Positive Affect Short Form

CONTACTS AND LOCATIONS:
Overall Officials: Alexia M Torke, MD, MS, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University Melvin & Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana